CLINICAL TRIAL: NCT01484808
Title: Retrospective Review of Reduce Data to Determine the Utility of PSADv While on Dutasteride for Predicting Prostate Cancer Incidence and Grade and Stage
Brief Title: The Utility of PSADv (PSA Density Velocity) While on Dutasteride for Predicting Prostate Cancer Incidence and Grade and Stage
Acronym: PSADv
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Urological Associates Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 8DUT115799
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-11

CONDITIONS: Prostate Cancer
Keywords: PSA Density; Prostate Cancer; Prostate Biopsy; PSA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a review of previously published data from a large prostate cancer prevention study known as REDUCE. It is the investigators intention to review whether prostate specific antigen (PSA) velocity (change over time) will predict the presence of prostate cancer and its grade and stage (severity).

DETAILED DESCRIPTION:
This is a review of previously published data from a large prostate cancer prevention study known as REDUCE that utilized a 5 ARI, dutasteride. It is the investigators intention to review whether PSA velocity (change over time) will predict the presence of prostate cancer and its grade and stage (severity) by two year biopsy. The investigator will review and compare data to a previously published study of similar design with finasteride.

ELIGIBILITY:
Inclusion Criteria:

* Men,
* 50-74 years old with elevated PSA (>=4) along with negative entry biopsy of the prostate who had a subsequent biopsy by 24 months.

Exclusion Criteria:

* Any positive biopsy of the prostate indicative of cancer upon entry

Ages: 50 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with PSA elevation (>=4), 50-74 years old with negative biopsy of the prostate at study entry
Sampling Method: Probability Sample
Enrollment: 6600 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven I Cohen, MD, Principal Investigator — University Urological Associates Inc.
Locations (1):
- Division of Urology, Brown University, Providence, Rhode Island, United States